CLINICAL TRIAL: NCT06813690
Title: Effects of Immediate and Delayed Repeated Cold Exposure After Physical Exertion: a Randomised Controlled Trial
Brief Title: Effects of Immediate and Delayed Repeated Cold Exposure After Physical Exertion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Applied Sciences and Arts of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Ron Clijsen, Prof. Dr., University of Applied Sciences and Arts of Southern Switzerland
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-D0116
Record Dates: First submitted 2025-01-20; First posted 2025-02-07 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Delayed Onset Muscle Soreness (DOMS); Inflammation; Muscle Pain; Muscle Damage
Keywords: Cold therapy for muscle recovery; Delayed Onset Muscle Soreness; Post-exercise recovery methods; Muscle pain and swelling reduction; Inflammation and recovery after exercise; Reducing exercise-induced muscle damage; Clinical trial on cryotherapy effectiveness
MeSH Terms: conditions — Inflammation; Myalgia | interventions — Cryotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A: Immediate Cooling (Experimental): In this group, cooling begins immediately after completing the muscle soreness protocol. Cooling is performed three times per day on the day of the protocol and continues for 72 hours. Both thighs are cooled using the "Cold Hot Maxi Pack" from Axanova for 20 minutes per session.
  Interventions: Device: Cold Therapy with Axanova Cold Hot Pearls Maxi Pack
- Group B: Delayed Cooling (Experimental): In this group, cooling begins 24 hours after completing the muscle soreness protocol. Cooling is also performed three times per day for 72 hours. Both thighs are cooled using the "Cold Hot Maxi Pack" from Axanova for 20 minutes per session.
  Interventions: Device: Cold Therapy with Axanova Cold Hot Pearls Maxi Pack
- Group C: Control Group (No Intervention): This group receives no cooling intervention or any other intervention after the muscle soreness protocol and throughout the study period.

INTERVENTIONS:
Device: Cold Therapy with Axanova Cold Hot Pearls Maxi Pack — This intervention involves the application of the Axanova Cold Hot Pearls Maxi Pack, a cooling device designed to provide targeted cold therapy. The device will be used to cool both thighs for 20-minute sessions, three times per day, following a muscle soreness protocol. The cold therapy aims to reduce inflammation, swelling, and muscle pain associated with Delayed Onset Muscle Soreness (DOMS). The intervention begins immediately after completing the muscle soreness protocol in Group A, and 24 hours later in Group B. Participants will receive cooling treatment for a total of 72 hours, with temperature and duration carefully monitored to ensure effective cooling.
  Arms: Group A: Immediate Cooling; Group B: Delayed Cooling

SUMMARY:
The goal of this clinical trial is to learn if applying cold therapy can reduce swelling, inflammation, and pain after physical activity in adults who experience muscle soreness (Delayed Onset Muscle Soreness, or DOMS). The main questions it aims to answer are:

* Can cold therapy reduce swelling and inflammation in muscles after exercise?
* Does cold therapy reduce muscle pain and discomfort (DOMS)?

Researchers will compare participants using the Axanova Cold Hot Pearls Maxi Pack to those not receiving any cold therapy to see if the cold application improves recovery outcomes.

Participants will:

* Perform physical activity designed to induce muscle soreness.
* Use the Axanova Cold Hot Pearls Maxi Pack on the affected area as directed.
* Report their level of muscle pain, stiffness, and swelling over the following 72 hours.

The study aims to provide new insights into the effectiveness of cold therapy for muscle recovery, focusing on pain relief, reduced swelling, and improved recovery time.

DETAILED DESCRIPTION:
Physical activity is influenced by factors such as the type, duration, and intensity. Depending on the extent of these factors and the associated recovery time, muscle damage, inflammation, and fatigue symptoms in the nervous system can occur. Additionally, energy substrate depletion and localized swelling may take place. Therefore, rapid recovery after intense exercise has become increasingly important. According to the meta-analysis by Bleakley et al. (2012), cold therapy is considered one of the most effective recovery methods after physical activity to delay Delayed Onset Muscle Soreness (DOMS).

DOMS consists of microscopic tears in muscle tissue, referred to as exercise-induced muscle damage, which can lead to delayed muscle soreness. DOMS typically peaks between 24 and 48 hours-sometimes up to 72 hours-after exercise and is characterized by muscle shortening, increased passive stiffness, swelling, reduced strength and performance, localized muscle soreness, and altered proprioception.

The physiological basis of cryotherapy lies in the removal of body heat through a reduction in tissue temperature. This results in decreased muscle pain perception, making the body feel more "awake" after training and reducing the sensation of fatigue. Additionally, cold exposure lowers heart rate and cardiac output while inducing vasoconstriction. The outcomes include smaller blood vessel diameters, reduced occurrence of edema, and improved oxygen supply to the cells. To maintain core body temperature, the central metabolism also increases, promoting the transport of metabolic waste products.

All these effects, in combination, may help reduce exercise-induced inflammation by minimizing the death or damage of hypoxic cells and reducing secondary tissue damage through decreased infiltration of leukocytes and monocytes (Bleakley et al. 2012, Hohenauer et al. 2015, Hubbard et al. 2004, Ostrowski et al. 2018).

ELIGIBILITY:
Inclusion Criteria

* Young, healthy adults aged between 18 and 30 years
* No surgical interventions on the musculoskeletal system in the trunk area or lower extremities

Exclusion Criteria

* Current pain conditions
* Current inflammatory conditions
* Medication use (excluding contraceptives)
* Pregnant participants
* Competitive athletes
* Children/teenagers
* Non-intact skin conditions (e.g., psoriasis)
* Known circulatory disorders
* Cold allergy (Raynaud's disease)

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 45 (Estimated)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in Muscle Pain (DOMS) | 72 hours
  Assessed using a visual analog scale (VAS) to measure self-reported muscle soreness in the thighs over 72 hours.
Reduction in Swelling | 72 hours
  Swelling of the anterior thigh muscles will be assessed using ultrasound diagnostics. A cross-sectional image of the thigh muscles will be captured, and the distance from the femur to the outer boundary of the muscle will be measured.
Inflammatory Marker Levels | 72 hours
  Blood samples will be taken in order for markers such as C-reactive protein (CRP) and creatine kinase (CK) levels to be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Ron Clijsen, Prof. Dr., Principal Investigator — University of Applied Sciences of Southern Switzerland
Locations (1):
- University of Applied Sciences and Arts of Southern Switzerland (SUPSI), Landquart, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Petrofsky JS, Khowailed IA, Lee H, Berk L, Bains GS, Akerkar S, Shah J, Al-Dabbak F, Laymon MS. Cold Vs. Heat After Exercise-Is There a Clear Winner for Muscle Soreness. J Strength Cond Res. 2015 Nov;29(11):3245-52. doi: 10.1519/JSC.0000000000001127. PMID 26502272
- [Background] Ostrowski J, Purchio A, Beck M, Leisinger J, Tucker M, Hurst S. Examination of Intramuscular and Skin Temperature Decreases Produced by the PowerPlay Intermittent Compression Cryotherapy. J Sport Rehabil. 2018 May 1;27(3):244-248. doi: 10.1123/jsr.2016-0244. Epub 2018 May 10. PMID 28422604
- [Background] Hubbard TJ, Denegar CR. Does Cryotherapy Improve Outcomes With Soft Tissue Injury? J Athl Train. 2004 Sep;39(3):278-279. PMID 15496998
- [Background] Hohenauer E, Taeymans J, Baeyens JP, Clarys P, Clijsen R. The Effect of Post-Exercise Cryotherapy on Recovery Characteristics: A Systematic Review and Meta-Analysis. PLoS One. 2015 Sep 28;10(9):e0139028. doi: 10.1371/journal.pone.0139028. eCollection 2015. PMID 26413718
- [Background] Bleakley C, McDonough S, Gardner E, Baxter GD, Hopkins JT, Davison GW. Cold-water immersion (cryotherapy) for preventing and treating muscle soreness after exercise. Cochrane Database Syst Rev. 2012 Feb 15;2012(2):CD008262. doi: 10.1002/14651858.CD008262.pub2. PMID 22336838

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-03-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT06813690/Prot_SAP_000.pdf